CLINICAL TRIAL: NCT01169610
Title: A 24-week Open-Label Feasibility Trial of Varenicline for Alcoholic Cigarette Smokers
Brief Title: Varenicline and Alcohol in Inpatient Addictions Program (IAP)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Frye, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-002699
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Alcoholism; Nicotine Dependence
Keywords: Alcohol; Smoking
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varenicline (Experimental)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline is an oral medication with a recommended dosage of 0.5 mg once daily for 3 days, increasing to 0.5 mg twice daily for days 4 to 7, and then to the maintenance dose of 1 mg twice daily for the remaining 23 weeks of treatment. All subjects will receive open-label varenicline in blister packs.
  Other Names: Chantix

SUMMARY:
The overall hypothesis of this line of research is that varenicline will decrease alcohol consumption and tobacco use and will increase alcohol and tobacco abstinence rates. In order to explore this hypothesis, the investigators will conduct a two-phase study: 1) an open label pilot study investigating the effect of varenicline on reduction of and abstinence from alcohol and tobacco; and 2) an optional MR spectroscopy to investigate whether glutamate and other brain metabolites correlate to measures of alcohol craving severity and/or subsequent varenicline treatment response.

DETAILED DESCRIPTION:
The goal of this proposal is to explore the potential efficacy of varenicline for reducing alcohol consumption among alcohol-dependent cigarette smokers. The hypothesis for the current study is that 24 weeks of varenicline will increase alcohol abstinence rates among smokers and decrease alcohol consumption among patients receiving inpatient addiction treatment for alcoholism. The investigators will also explore whether varenicline has a beneficial effect on tobacco abstinence rates in this population of tobacco users.

The investigators will conduct an open-label pilot study to determine clinical efficacy and employ neuroimaging techniques to evaluate how glutamate and other brain metabolites correlate to measures of alcohol craving severity and/or subsequent varenicline treatment response. The investigators will enroll 20 subjects receiving treatment in the Mayo Clinic Inpatient Addictions Program (IAP) and compare outcomes with patients participating in a similar 6-month open-label study of acamprosate.

The Primary aims of this study are:

1. To obtain preliminary evidence of efficacy of varenicline (0.5 mg once daily for 3 days, 0.5 mg twice daily for days 4-7, 1 mg twice a day for remaining 23 weeks) for increasing continuous alcohol abstinence rates at 3 and 6 months among patients with alcohol and tobacco dependence who have completed treatment at the Mayo Clinic IAP.
2. To obtain preliminary evidence of efficacy of varenicline (0.5 mg once daily for 3 days, 0.5 mg twice daily for days 4-7, 1 mg twice a day for remaining 23 weeks) for decreasing the number of heavy drinking days (> 5 drinks/day for men and > 4 drink/day for women) at 3 and 6 months among patients with alcohol and tobacco dependence who have completed treatment at the Mayo Clinic IAP.
3. To obtain preliminary data on baseline and baseline to endpoint change in CSF volume corrected concentrations of the dorsal striatal glutamate, glutamate + glutamine, and NAA measures through MR spectroscopy before and after 30 days of varenicline treatment among patients with alcohol and tobacco dependence who have completed treatment at the Mayo Clinic IAP.

Secondary aims:

1. To obtain preliminary evidence of efficacy of varenicline (0.5 mg once daily for 3 days, 0.5 mg twice daily for days 4-7, 1 mg twice a day for remaining 23 weeks) for increasing the 7-day point prevalence smoking abstinence rates and prolonged smoking abstinence at 3 and 6 months among patients with alcohol and tobacco dependence who have completed treatment at the Mayo Clinic IAP.
2. To assess the tolerability of varenicline (0.5 mg once daily for 3 days, 0.5 mg twice daily for days 4-7, 1 mg twice a day for remaining 23 weeks).

ELIGIBILITY:
Subjects will be eligible for enrollment if they:

1. Are > 18 and < 70 years of age
2. Are admitted to the inpatient addiction program (IAP) in the Generose Building at Saint Marys Hospital
3. Have been diagnosed with alcohol dependence based on DSM-IV-TR criteria and confirmed by Psychiatric Research Interview for Substance and Mental Disorders (PRISM)
4. Smoke at least 10 cigarettes/day for ≥ 6 months
5. Are able to participate fully in all aspects of the study
6. Have been provided with, understand, and have signed the informed consent; and
7. Agree to identify collateral individuals for contact purposes to facilitate follow-up appointments.

Patients will be excluded from participation if they:

1. Meet DSM-IV criteria of schizophrenia or other non-affective psychotic disorder
2. Have had psychotic symptoms within the past month
3. Have an Axis I disorder requiring new pharmacotherapy
4. Have a predominant Axis II disorder
5. Have used an investigational drug within 30 days of enrollment
6. Have started Naltrexone or Acamprosate during this same IAP admission
7. Have a history (past 3 months) of drug abuse (excluding caffeine and marijuana)
8. Have active suicidality as measured by screening questions from the Columbia-Suicide Severity Rating Scale (C-SSRS), (Posner 2008) outlined below:

   a. "Yes" response to questions 1, 2, or 3 with significant intensity level endorsed as: i. Frequency: score of 4 or 5 ii. Duration: score of 3, 4 or 5 iii. Controllability: score of 0, 4, or 5 iv. Deterrents: score of 0, 4 or 5 v. Reasons for Ideation: score of 1, 2, 3, 4 or 5 b. "Yes" response to question 4 c. "Yes" response to question 5
9. Have a history of medically serious suicide attempt within 5 years
10. Have a history of any major cardiovascular events including arrhythmias, congestive heart failure, unstable angina, acute MI or coronary angioplasty
11. Are pregnant, lactating, or of child bearing potential, likely to become pregnant during the medication phase and not willing to use a reliable form of contraception. Reliable forms of contraception include diaphragm or condom (with spermicidal), injections, intrauterine device [IUD], surgical sterilization and abstinence;
12. Have clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, respiratory or metabolic disease
13. Have another household member or relative participating in the study
14. Have a known allergy to varenicline
15. Are individuals, in the investigators opinion, unable to comply with study procedures
16. Are unable to provide written informed consent in English
17. Are on hemodialysis or have a history of kidney disease.

Patients will be excluded from participation in the MR spectroscopy portion of the study if they have:

1. Claustrophobia
2. A history of major head trauma with loss of consciousness > 5 minutes or skull fracture
3. A history of previous neurological event (e.g., epilepsy, stroke, transient ischemic attack)
4. Implanted metal objects (e.g., pacemakers; aneurysm clips; metal prostheses, joints, rods, or plates)
5. Contraindication to MRI scanning.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 1/2011 - 9/2012
Groups:
- Open Label: Varenicline : Varenicline is an oral medication with a recommended dosage of 0.5 mg once daily for 3 days, increasing to 0.5 mg twice daily for days 4 to 7, and then to the maintenance dose of 1 mg twice daily for the remaining 23 weeks of treatment. All subjects will receive open-label varenicline in blister packs.
Period: Overall Study
Arm/Group | Open Label
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: data not analyzed for 1 participant enrolled
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Continuous Alcohol Abstinence
Description: No consumption of alcohol (not even a single drink) during the specified interval of time. This will be a self-reported outcome.
Time Frame: Two years
Population: Data not analyzed for 1 participant enrolled
Arm/Group | Open Label
Number analyzed (Participants) | 0

2. Primary Outcome: Heavy Drinking Days
Description: Number of drinking days > 5 drinks/day for men and > 4 drink/day for women. This will be a self-reported outcome.
Time Frame: Two years
Population: data not analyzed for 1 participant enrolled
Arm/Group | Open Label
Number analyzed (Participants) | 0

3. Secondary Outcome: 7-day Point Prevalence Smoking Abstinence
Description: Negative response to the question, "Have you used any type of tobacco, even a puff, in the past 7 days." This will be a self-reported outcome biochemically-confirmed with exhaled-air carbon monoxide (CO) < 8 parts per million (ppm) during the medication phase.
Time Frame: Two years
Population: data not analyzed for 1 participant enrolled
Arm/Group | Open Label
Number analyzed (Participants) | 0

4. Secondary Outcome: Prolonged Smoking Abstinence
Description: Self-reported all tobacco abstinence since two weeks after target quit date (TQD) which will be during their 28-day stay in the IAP on day 8 of varenicline therapy. Negative response to the question, "Have you used any type of tobacco, even a puff, for 7 consecutive days or at least once each week on two consecutive weeks since xx/xx/xxxx?" Note: xx/xx/xxxx corresponds to the date two weeks after the target quit date (TQD).
  Biochemically-confirmed abstinence at the visit for which prolonged abstinence is being obtained.
Time Frame: Two years
Population: data not analyzed for 1 participant enrolled
Arm/Group | Open Label
Number analyzed (Participants) | 0

5. Secondary Outcome: Tolerability of Varenicline
Description: Tolerability will be defined by the number of adverse events experienced by patients.
Time Frame: Two years
Population: data not analyzed for 1 participant enrolled
Arm/Group | Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes